CLINICAL TRIAL: NCT05820646
Title: Effect of Boswellia Sacra Versus Calcium Hydroxide as an Intracanal Medicament on Postoperative Pain Intensity and Bacterial Load Reduction in Necrotic Mandibular Premolars: A Randomized Clinical Trial
Brief Title: Effect of Boswellia Sacra as an Intracanal Medicament on Postoperative Pain Intensity and Bacterial Load Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Helmy Abd-Elghafar Abo Kashwa, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3.7.1
Record Dates: First submitted 2023-03-28; First posted 2023-04-19 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Intervention
MeSH Terms: interventions — Frankincense

STUDY DESIGN:
Intervention Model Description: Parallel randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors (patients, microbiologist and statistician) will not know Which group the participants will be related to?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with necrotic mandibular premolars will be treated with boswellia sacra (Experimental): 25-45 years old patients with necrotic single rooted mandibular premolar with single canal with periapical lesion will be treated with boswellia sacra as an intracanal medicament for 3 days
  Interventions: Other: Boswellia Sacra
- Patient with necrotic mandibular premolar will be treated with boswellia sacra (Experimental): 25-45 years old patients with necrotic single rooted mandibular premolar with single canal with periapical lesion will be treated with boswellia sacra as an intracanal medicament for 7 days
  Interventions: Other: Boswellia Sacra
- Patients with necrotic mandibular premolar will be treated with calcium hydroxide (Active Comparator): 25-45 years old patients with necrotic single rooted mandibular premolar with single canal with periapical lesion will be treated with calcium hydroxide as an intracanal medicament for 7 days
  Interventions: Other: Boswellia Sacra

INTERVENTIONS:
Other: Boswellia Sacra — 1. Boswellia Sacra used as an intracanal medicament for 3 days
  2. Boswellia Sacra used as an intracanal medicament for 7 days

SUMMARY:
This research will study the effect of Boswellia Sacra versus calcium hydroxide as an intracanal medicament on postoperative pain intensity measured using numerical rating scale (NRS) and bacterial load reduction reduction determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml) in mandibular premolars with necrotic pulp.

DETAILED DESCRIPTION:
Primary outcome Postoperative pain measured using numerical rating scale (NRS)

1. After placement of intracanal medicament at 6, 12, 24 and 48 hours.
2. After root canal obturation at 6, 12, 24 and 48 hours.

Secondary outcomes Bacterial load reduction determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml) .

1. Sample 1 (S1): after access preparation and pre-instrumentation.
2. Sample 2 (S2): post-instrumentation.
3. Sample 3 (S3): post-intracanal medicament removal at 3 or 7 days according to the group.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25-45 years old.
2. Males or females.
3. Healthy patients whom are categorized as I or II according to The American Society of Anesthesiologists. (ASA I or II)
4. Patients' accepting to participate in the trial.
5. Patients who can understand pain scale and can sign the informed consent.
6. Mandibular Single rooted premolars, having single root canal:

   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pulpal pain.
   * Positive pain on percussion denoting apical periodontitis.
   * Periapical radiolucency not exceeding 2*2 mm radiographically.
   * Normal occlusal contact with opposing teeth.

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders (ASA III or IV).
2. If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively as it might alter their pain perception.
3. Pregnant women: to avoid radiation exposure, anesthesia, medication and hormonal Fluctuation that might increase pain prevalence.
4. Patients reporting bruxism, clenching, TMJ problems or traumatic occlusion: to avoid further pressure on inflamed tooth which induce subsequent irritation and inflammation.
5. Patients with two or more adjacent teeth requiring endodontic treatment.
6. Teeth that requires further procedural steps or multidisciplinary approach, which is out of this experiment's scope:

   i. Association with swelling or fistulous tract. ii. Acute periapical abscess. iii. Mobility Grade II or III. iv. Pocket depth more than 5mm. v. Previous root canal treatment. vi. Non -restorable vii. Immature roots viii. Radiographic evidence of external or internal root resorption, vertical root fracture, perforation, calcification.
7. Inability to perceive the given instructions.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured using numerical rating scale | 48 hours.
  postoperative pain will be recorded after placement of intracanal medicament and after root canal obturation using numerical rating scale ,An 11-point scale from 0-10 representing pain intensity ,"10" being the most intense pain conceivable.

SECONDARY OUTCOMES:
Bacterial load reduction | T0=Baseline immediate after access preparation . T1=Post-instrumentation. T3=post-intracanal medicament removal at 3 or 7 days according to the group.
  Bacterial load reduction determined by bacterial counting using agar culture technique after root canal preparation (Number of colony forming unit per millilitre)
Incidence of inter-appointment swelling | Up to 48 hours post- operatively
  • Incidence of inter-appointment swelling measured using visual analog scale of postoperative swelling (VAS)
Incidence of analgesic intake after root canal treatment | Up to 48 hours post- operatively
  Incidence of analgesic intake after root canal treatment, using numerical counting.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A. El.Baz, Study Director — Professor
Locations (1):
- Cairo University Hospital ,Endodontic clinic, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No